CLINICAL TRIAL: NCT04942158
Title: Efficacy of Non-instrumentation Endodontic Treatment With an Antibiotic Mix Paste in Primary Molars: a Multicenter Randomized Clinical Trial With 2 Years of Follow-up
Brief Title: Non-instrumentation Root Canal Treatment of Primary Molars
Acronym: EndoDecide-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Santa Catarina Federal University (Other); Rio de Janeiro State University (Other); Iguaçu University (Unknown)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDODECIDE-001
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Dental Pulp Diseases; Dental Pulp Necrosis
Keywords: Endodontic treatment; Primary teeth; Non-instrumentation technique; CTZ paste; Pulpectomy
MeSH Terms: conditions — Dental Pulp Diseases; Dental Pulp Necrosis | interventions — Zinc Oxide

STUDY DESIGN:
Intervention Model Description: Multi-center, open label, non-inferiority randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTZ group (Experimental): Non-instrumentation endodontic treatment and use of a paste containing two antibiotics (chloramphenicol and tetracycline) and zinc oxide and eugenol (CTZ paste)
  Interventions: Procedure: Non-instrumentation technique with use of CTZ paste
- ZOE group (Active Comparator): Endodontic treatment with instrumentation and filling with Zinc Oxide and Eugenol paste (ZOE paste)
  Interventions: Procedure: Instrumentation technique and filling with Zinc Oxide and Eugenol paste

INTERVENTIONS:
Procedure: Non-instrumentation technique with use of CTZ paste — After local anesthesia and rubber dam isolation, the pulp chamber will be accessed. After the location of root canals entrance, an initial irrigation will be conducted using 1% sodium hypochlorite. Then, a paste containing two antibiotics (chloramphenicol and tetracycline) and zinc oxide and eugenol (CTZ paste) will be placed in the pulp chamber floor, into the root canal entrances. Then, a layer of glass ionomer cement will be placed, and the teeth will be restored with bulk-fil resin composite.
  Arms: CTZ group
Procedure: Instrumentation technique and filling with Zinc Oxide and Eugenol paste — After anesthesia and rubber dam isolation, pulp chamber will be accessed with burs, and the root canals entrance will be prepared using a Gates Glidden bur. The root canal length determination will be done subtracting 1 mm from the radiographic measurements performed on the different roots. The instrumentation will be performed with 21mm stainless steel endodontic hand K-files, with International Organization for Standardization (ISO) tip ranging from #08 to #35. Irrigation will be performed using 1% sodium hypochlorite. After the last file, a final irrigation will be conducted with ethylenediaminetetraacetic acid and tegentol (EDTA-T) and 0.9% sodium chloride solution, and the root canals will be dried with paper points. Then, the root canals will be filled with a Zinc Oxide and Eugenol paste (ZOE paste), inserted into the root canals with a lentulo spiral. A layer of glass ionomer cement will be placed, and the teeth will be restored with bulk-fil resin composite.
  Arms: ZOE group

SUMMARY:
This randomized clinical trial intended to evaluate the efficacy of a technique of root canal treatment of deciduous molars with non-instrumentation of root canals and use of a paste containing antibiotics (chloramphenicol and tetracycline) and zinc oxide and eugenol (CTZ group). The hypothesis is that the efficacy of non-instrumentation treatment is non-inferior than the standard treatment involving manual instrumentation of root canals and filling with zinc oxide and eugenol paste (ZOE group) after 24 months of follow-up. Children will be randomly allocated to one of the two groups: CTZ group or ZOE group. In the CTZ group, after the location of root canals entrance, an initial irrigation will be conducted using 1% sodium hypochlorite. Then, CTZ paste will be placed in the pulp chamber floor, over the root canal entrances. The instrumentation of the root canals will not be performed for children allocated to this group. For the ZOE group, manual instrumentation with endodontic K files will be performed, aided by irrigation with 1% sodium hypochlorite. After the end of the instrumentation, root canals will be filled with ZOE paste. All teeth will be restored with bulk-fil resin composite. Children will be followed-up for 6, 12, 18 and 24 months after the treatment. The primary endpoint will be the success of endodontic treatment evaluated by clinical and radiographic methods after 24 months. Based on a non-inferiority limit of 15% in the success rate, an anticipated sample size of 218 (109 per group) was estimated, divided among the centers. This sample size was further corrected two times (due to slower-than-anticipated recruitment, and due to the drop of a center participant of the study), reaching a required minimum sample size of 182 participants (91 participants per group).

Other secondary endpoints will be clinical time spent with the treatments, children's behavior during the treatment, discomfort immediately after the end of the treatment reported by the children, post-operative pain, improvement in the negative impact of Oral Health-Related Quality of Life, costs and cost-efficacy.

DETAILED DESCRIPTION:
Most techniques for endodontic treatment in primary teeth require instrumentation of root canals and filling with an absorbable paste. This filling material could be pastes based on zinc oxide and eugenol, calcium hydroxide or iodoform, or filling materials composed by mixture of some of these components. This method, however, requires a long clinical time, which can be a challenge in the Pediatric Dentistry clinical practice. Therefore, some alternative techniques in which non-instrumentation is necessary have been purposed.

The non-instrumentation technique most used in Brazil is a technique previously described, in 1964. This method involves the access to pulp chamber and removal of necrotic tissue with irrigation. After that, with no instrumentation of the root canals, a medicament containing zinc oxide and eugenol and two antibiotics, chloramphenicol and tetracycline, is placed in the entrance of the canals, and the restoration of the teeth is performed. Although the non-instrumentation methods for endodontic treatment of primary teeth are attractive and demand a short clinical time, strong evidence from well-conducted clinical trial lacks.

Therefore, this four-center parallel-arms non-inferiority randomized clinical trial was designed to evaluate the efficacy of a non-instrumentation of root canals and use of a paste containing antibiotics (chloramphenicol and tetracycline) and zinc oxide and eugenol (CTZ) technique for endodontic treatment of primary molars. The hypothesis is that the efficacy of non-instrumentation treatment is non-inferior to the standard treatment involving manual instrumentation of root canals and filling with zinc oxide and eugenol (ZOE) paste after 24 months of follow-up. Children who look for dental treatment in one of four participating centers and who have at least one primary molar requiring endodontic treatment will be eligible. If the child has more than one molar with pulp involvement, the included tooth will be determined by chance. Other teeth will be treated, but they will not be included in the study. The participating centers are the dental schools of Santa Catarina Federal University, University of Sao Paulo, Rio de Janeiro State University and Iguaçu University. Included children will be randomly allocated to one of the two groups (allocation ratio of 1:1): CTZ group (non-instrumentation technique) and ZOE group (standard treatment).

Randomization list will be generated in an appropriate website (www.sealedenvelopes.com), in permuted blocks (2, 4, and 8 samples) and stratified for the center. The sequence will be enclosed in individual opaque envelopes separated by the stratum. The disclosure of the allocated group will occur when the children will be seated in the dental chair, after the anesthesia, rubber dam isolation and opening of the tooth included for that child. Than the included tooth will be allocated to the CTZ group or to ZOE group. After the treatment, children will be followed-up for 6, 12, 18 and 24 months. Evidence of treatment failure in any period will be recorded, and the teeth will be extracted.

The primary endpoint will be the success of the dental treatment after 24 months of follow-up (teeth with no evidence of failure in all follow-ups). The sample size calculation was estimated based on a success rate of 92% obtained in pulpectomies using ZOE from a previous systematic review (Coll et al., 2020), a non-inferiority limit of 15%, a significance level of 5% and statistical power of 90%. It was added 20% to this number to contemplate possible drop-outs and 60% due to the multi-center design. The anticipated sample size was 218 teeth (109 per group), divided among the centers.

However, in March 2023, we decided to modify the original sample size from 218 to 200 participants, due to slower-than-anticipated recruitment. With this sample, considering the same parameters, we maintained a statistical power of around 90% (90.6%).

Another problem we have noticed in the last year (between March 2024 and March 2025) is that one of the study centers (Iguaçu University) was unable to include and follow up an adequate number of participants (less than 10 children in almost two years). Therefore, we decided to drop this center, and we recalculated the sample size, adjusting the correction for the multicenter design to 1.4. Our final minimum sample size to reach an adequate power, considering the prespecified parameters - 5% of significance level, 90% of statistical power, 92% of success rate for the control group, a non-inferiority limit of 15% and adding 60% to this number (20% for drop-outs and 40% due to multicenter design) - was 182 participants. As our randomization process was stratified per center, we do not expect a significant bias due to the center drop.

Masking will not be possible for participants, operators, researchers, or even outcome assessors due to the different nature of the treatments. However, the outcome assessor will not be informed of the allocated group for each tooth.

Other secondary endpoints will be the clinical time spent with the treatments, children's behavior during the treatment, discomfort immediately after the end of the treatment reported by the children, post-operative pain, short- and long-term improvement in the negative impact of Oral Health-Related Quality of Life, costs and cost-efficacy. The frequency of treatment success after 24 months will be compared between the groups in the intention-to-treat population considering the non-inferiority limit of 15% by the Miettinen-Nurminen's method. Sensitivity analysis will be conducted through non-inferiority Cox regression. For this, the period that the treatment failure occurred will be recorded. Secondary outcomes will be compared by proper statistical tests considering two-tailed hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Children who look for dental treatment
* Children with at least one primary molar with clinical and/or radiographic signs of pulpal involvement
* Formal consent of the children's parents or legal guardians agreeing with the participation of the children
* Write or verbal assent of the children in participating of the study

Exclusion Criteria:

* Children with special needs
* Children with report of allergy to the medications used in the pastes
* Children with a negative behavior in the inclusion session

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Success of endodontic treatment | 24 months
  The success of the endodontic treatment is a dichotomous variable that will be defined through clinical and radiographic evaluation after 24 months. Clinical criteria for determining success will be the absence of fistula, edema, pain, pathological mobility, presence of periodontal health or physiological primary molar exfoliation. Radiographic signs of success will be: absence of bone rarefaction, or in the presence of previous endodontic lesion, reduction or non-evolution of this lesion, compatible root resorption with the eruptive phase, absence of pathological root resorption and presence of restorative material isolating the filling paste from the oral cavity. In the presence of any signs of failure in any period of follow-up, the treatment will be considered unsuccessful. The main comparisons between the groups will be done considering the frequency rate of success treatment 24 months after the treatment, when absence of failure was detected in all follow-ups.

SECONDARY OUTCOMES:
Clinical time | During the treatment procedure
  The clinical operating time from the topical anesthesia to the removal of the rubber dam isolation after tooth restoration will be recorded with a digital chronometer by the dental assistant. The average time (quantitative variable) will be compared between the groups.
Children's behavior during the treatment | During the treatment procedure
  This outcome will be assessed during the treatment by an external researcher using the Frankl Scale, an ordinal scale classifying the behavior during the treatment with four categories varying from definitely negative behavior (score 1) to definitely positive behavior (score 4). This assessor will classify the children's behavior in the period between the topical anesthesia until to the removal of rubber dam isolation. This endpoint will be considered as a qualitative ordinal variable.
Children's discomfort immediately after the intervention | Immediately after intervention
  This variable will be reported by the participant using the Facial Image Scale, immediately after the end of the endodontic intervention. This is an ordinal scale with five representative faces ranging from a very sad and crying face (score 5) from a very happy and smiley face (score 1). Immediately after the end of the treatment, an external assessor will show the scale for the children and will ask: "Which of these faces reflects how you feel after treating your tooth?". The score related to the face that children indicated will be recorded. The outcome will be summarized and compared as a qualitative ordinal variable.
Postoperative pain, edema or fistula | Two days after the end of the intervention
  Two days after the endodontic treatment, the operator will make a phone call to the children's parents. The occurrence of postoperative pain will be evaluated through 3 questions that will be done by the assessor: Has your kid reported pain in the treated teeth (yes or no)? Has you noticed some edema (swelling) or fistula with pus (yes or no)?; and Did your kid need of analgesic medication intake (yes or no)?. These variables will be compared separately between the groups as dichotomous variables.
Short-term impact of the treatment on Oral Health-Related Quality of Life reported by the children | One week after the end of the intervention
  This outcome will be evaluated considering the scores obtained through a questionnaire to assess the Oral Health-Related Quality of Life (OHRQoL) answered by the children. The instrument that will be applied is the short-form of the Child Perceptions Questionnaire for children from 8 to 10 years old (CPQ 8-10) at the baseline, after the inclusion of the children (before the disclosure of the allocated group). The instrument has 16 questions, and five answer options are given for each question. A score ranging from 0 to 4 is given for each question, and the final score is obtained by the sum of all items. The higher the score obtained, the worse the OHRQoL. After 1 week of the end of the treatment, a new questionnaire will be applied. The mean of change scores and the effect sizes considering these two questionnaires will be compared between the groups.
Long-term impact of the treatment on Oral Health-Related Quality of Life reported by the children | 24 months
  In the 24 months follow-up period, a children will answer again the short version of the CPQ 8-10. The mean of change scores and the effect sizes considering these answers and the scores obtained with the instrument applied at the baseline will be compared between the groups.
Short-term impact of the treatment on Oral Health-Related Quality of Life reported by the parents | One week after the end of the intervention
  This outcome will be evaluated considering the scores obtained through a questionnaire to assess the Children's Oral Health-Related Quality of Life (OHRQoL), using the answers by the parents as proxy. The instrument that will be applied is the Early Childhood Oral Health Impact Scale (ECOHIS) at the baseline, after the inclusion of the children (before the disclosure of the allocated group). The instrument has 13 questions, and six answer options are given for each question. A score ranging from 0 to 5 is given for each question, and the final score is obtained by the sum of all items. The higher the score obtained, the worse the OHRQoL. After 1 week of the end of the treatment, a new questionnaire will be applied. The mean of change scores and the effect sizes considering these two questionnaires will be compared between the groups.
Long-term impact of the treatment on Oral Health-Related Quality of Life reported by the parents | 24 months
  In the 24 months follow-up period, the children's guardian who responded the ECOHIS at the baseline and one week after the intervention will answer again the ECOHIS. The mean of change scores and the effect sizes considering these answers and the scores obtained with the instrument applied at the baseline will be compared between the groups.
Costs | Immediately after intervention
  Costs of each procedure, with no considering the follow-up evaluations or failures, will be calculated per each tooth treated. In children with more than one tooth treated, the values will be multiplied by the number of treated teeth.
Cost-efficacy | 24 months
  The costs of each treatment will be added to the cost of the failures and will be adjusted by the efficacy obtained with each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto M Mendes, PhD, Principal Investigator — University of Sao Paulo
Locations (4):
- Brazil (4):
  - Iguaçu University, Itaperuna, Rio de Janeiro
  - Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro
  - Santa Catarina Federal University, Florianópolis, Santa Catarina
  - School of Dentistry, University of Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
The anonymous Individual Participating Data (IPD) containing baseline characteristics of the children and the teeth included, and results obtained for all primary and secondary endpoints, including appropriate dictionaries for the data will be shared in an institutional public repository of data after the acceptance of the manuscript containing the analysis of the primary endpoint (about 3 years after the inclusion of the first participant). The data will be shared as Excel Spreadsheet Format. The repository is the Institutional repository of scientific data of the University of São Paulo (repositorio.uspdigital.usp.br/) We will also share the descriptions of the Standard Operating Procedures created for two treatment groups as a text file, after the finish of the inclusions of the participants.
Time Frame: After the acceptance of the manuscript containing the main analysis of the primary outcome (about 3 years after the beginning of the study).
Access Criteria: The access will be allowed for any researcher. Utilization of the data should be done with adequate citation of the original source.
URL: http://repositorio.uspdigital.usp.br/

REFERENCES:
- [Background] Coll JA, Dhar V, Vargas K, Chen CY, Crystal YO, AlShamali S, Marghalani AA. Use of Non-Vital Pulp Therapies in Primary Teeth. Pediatr Dent. 2020 Sep 15;42(5):337-349. PMID 33087217
- [Background] Pezzini Soares J, Cardoso M, Bolan M. Demystifying behaviour and dental anxiety in schoolchildren during endodontic treatment for primary teeth-controlled clinical trial. Int J Paediatr Dent. 2019 May;29(3):249-256. doi: 10.1111/ipd.12468. Epub 2019 Feb 1. PMID 30656782
- [Background] Duarte ML, Pires PM, Ferreira DM, Pintor AVB, de Almeida Neves A, Maia LC, Primo LG. Is there evidence for the use of lesion sterilization and tissue repair therapy in the endodontic treatment of primary teeth? A systematic review and meta-analyses. Clin Oral Investig. 2020 Sep;24(9):2959-2972. doi: 10.1007/s00784-020-03415-0. Epub 2020 Jul 14. PMID 32666347
- [Background] Cappiello J. Pulp treatment in primary incisors [Spanish]. Rev Asoc Odontol Argent. 1964; 52(4): 139-145.
- [Background] de Deus Moura Lde F, de Lima Mde D, Lima CC, Machado JI, de Moura MS, de Carvalho PV. Endodontic Treatment of Primary Molars with Antibiotic Paste: A Report of 38 Cases. J Clin Pediatr Dent. 2016;40(3):175-7. doi: 10.17796/1053-4628-40.3.175. PMID 27472562